CLINICAL TRIAL: NCT06529263
Title: The Effect of Newborn Massage on Comfort Level and Vital Signs
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, aysel kokcudogan, Ph.D., Asst. Prof., Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-10840098-772.02-7436
Record Dates: First submitted 2024-07-18; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Newborn
Keywords: Newborn; infant massage; vital signs; comfort

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage group (Experimental): is the newborn massage group.The experimental group was massaged twice a day for 15 minutes 30 minutes after feeding and routine care for 4 days.
  Interventions: Other: newborn massage
- Control group (No Intervention): is the group without intervention

INTERVENTIONS:
Other: newborn massage — Newborn massage is one of the complementary treatment methods that support the treatment and contribute to the development of the baby
  Arms: Massage group

SUMMARY:
This study was planned as a randomized, controlled, experimental study to examine the effect of neonatal massage on the comfort level and vital signs of newborn babies.An answer to the question "Does massage applied to infants in the neonatal period have an effect on vital signs and comfort level?" will be sought.

DETAILED DESCRIPTION:
The sample of the study consisted of a total of 60 infants, 30 in the experimental group and 30 in the control group, who were hospitalized in the Neonatal Intensive Care Unit of a City Hospital between December 2022 and April 2023, whose parents' written and verbal consent was obtained for participation in the study after being informed, and who met the inclusion criteria. "Data Collection Form", 'Life Findings Assessment Form' and 'Newborn Comfort Behaviors Scale' prepared by the researchers were used as data collection tools. Newborns in the experimental group were massaged twice a day for 15 minutes 30 minutes after feeding and routine care for 4 days. The data obtained in the study will be analyzed using SPSS (Statistical Package for Social Sciences) for Windows 22.0 program.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 37-42 weeks,
* Birth weight of 2500 grams and above,
* The infant was hospitalized in the Neonatal Intensive Care Unit during data collection,
* Completion of 24 hours after birth

Exclusion Criteria:

* Gestational age below 37 weeks,
* Birth weight below 2500 grams,
* Refusal of the parent to participate in the study,
* The baby is on mechanical ventilation

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Body temperature | Measurements were taken before and after the newborn massage 2 times a day for 4 days.
  Measurements were taken at 10.00 am in the morning. After 30 minutes, neonatal massage was performed. The newborn massage lasted 15 minutes. Measurements were taken again 30 minutes after the massage. Measurements were taken at 22.00 in the evening. Newborn massage lasted 15 minutes. Measurements were taken again 30 minutes after the massage was finished (Measurements were taken before and after the massage performed 2 times a day).
Pulse | Measurements were taken before and after the newborn massage 2 times a day for 4 days.
  Measurements were taken at 10.00 am in the morning. After 30 minutes, neonatal massage was performed. The newborn massage lasted 15 minutes. Measurements were taken again 30 minutes after the massage. Measurements were taken at 22.00 in the evening. Newborn massage lasted 15 minutes. Measurements were taken again 30 minutes after the massage was finished (Measurements were taken before and after the massage performed 2 times a day).
Respiration | Measurements were taken before and after the newborn massage 2 times a day for 4 days.
  Measurements were taken at 10.00 am in the morning. After 30 minutes, neonatal massage was performed. The newborn massage lasted 15 minutes. Measurements were taken again 30 minutes after the massage. Measurements were taken at 22.00 in the evening. Newborn massage lasted 15 minutes. Measurements were taken again 30 minutes after the massage was finished (Measurements were taken before and after the massage performed 2 times a day).
Understanding Pulse Oximetry | Measurements were taken before and after the newborn massage 2 times a day for 4 days.
  Measurements were taken at 10.00 am in the morning. After 30 minutes, neonatal massage was performed. The newborn massage lasted 15 minutes. Measurements were taken again 30 minutes after the massage. Measurements were taken at 22.00 in the evening. Newborn massage lasted 15 minutes. Measurements were taken again 30 minutes after the massage was finished (Measurements were taken before and after the massage performed 2 times a day).
Newborn comfort behaviors scale | Measurements were taken before and after the newborn massage 2 times a day for 4 days.
  Measurements were taken at 10.00 am in the morning. After 30 minutes, neonatal massage was performed. The newborn massage lasted 15 minutes. Measurements were taken again 30 minutes after the massage. Measurements were taken at 22.00 in the evening. Newborn massage lasted 15 minutes. Measurements were taken again 30 minutes after the massage was finished (Measurements were taken before and after the massage performed 2 times a day).
  The comfort levels of newborn babies before and after massage were checked. Evaluation was made using the neonatal comfort scale. The lowest score that can be obtained from the Neonatal Comfort Behavior Scale is 6 and the highest score is 30. If the total score of the scale is between 14-30, it is emphasized that the baby has pain or distress, the baby is uncomfortable and needs interventions to provide comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Kokcu Dogan, Study Director — Faculty Member
Locations (1):
- Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No